CLINICAL TRIAL: NCT00776230
Title: Immunogenicity of a Commercial Batch of the Japanese Encephalitis Vaccine IC51 up to Twenty-four Months Post Filling. An Open-label, Multicenter, Phase 3 Study
Brief Title: Immunogenicity of a Commercial Batch of JEV IC51 up to 24 Months Post Filling
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IC51-314
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Results first posted 2014-01-23 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-03

CONDITIONS: Japanese Encephalitis
MeSH Terms: conditions — Encephalitis, Japanese | interventions — Japanese Encephalitis Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IC51 (~12 months post filling) (Active Comparator): 6 mcg (~12 months post filling)
  Interventions: Biological: IC51
- IC51 (~18 months post filling) (Active Comparator): 6 mcg (~18 months post filling)
  Interventions: Biological: IC51
- IC51 (~24 months post filling) (Active Comparator): 6 mcg (~24 months post filling)
  Interventions: Biological: IC51

INTERVENTIONS:
Biological: IC51 — 6 mcg im. at day 0 and day 28
  Other Names: Japanese Encephalitis vaccine

SUMMARY:
The objective is to assess immunogenicity of a commercial IC51 batch at 3 different time points post filling (12, 18, 24 months) in terms of Geometric Mean Titers (GMT) for anti-JEV neutralizing antibodies at Day 56 after the first vaccination.

DETAILED DESCRIPTION:
Open-label, multicenter, phase 3 study assessing immunogenicity at various time points throughout the shelf-life of a commercial batch of IC51 (Batch IC51/07F/008) The study population consists of male and female healthy subjects, aged at least 18 years.

The study will be performed at 3 study centers in Germany and Austria. Three sequential cohorts, each containing 100 subjects, will be enrolled into the study at approximately 12, 18 and 24 months after filling of the commercial batch IC51/07F/008 of IC51

ELIGIBILITY:
Inclusion Criteria:

* Male and female healthy adults aged at least 18 years with written informed consent and either no childbearing potential or negative pregnancy test.

Exclusion Criteria:

* History of immunodeficiency or immunosuppressive therapy, known HIV infection, drug addiction including alcohol dependence, prior vaccination against JE

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Hatzenbichler, Study Director — Valneva Austria GmbH
Locations (3):
- Zentrum für Reisemedizin, Vienna, Vienna, Austria
- Germany (2):
  - Universitätsklinikum Rostock, Rostock, Rostock
  - Berliner Zentrum Reise- und Tropenmedizin, Berlin, State of Berlin

RESULTS

PARTICIPANT FLOW:
Groups:
- IC51 Cohort 1: vaccinations with IC51 6 mcg i.m. on Day 0 and Day 28; batch age: ~12 months after filling;
- IC51 Cohort 2: vaccinations with IC51 6 mcg i.m. on Day 0 and Day 28; batch age: ~18 months after filling;
- IC51 Cohort 3: vaccinations with IC51 6 mcg i.m. on Day 0 and Day 28; batch age: ~24 months after filling;
Period: Overall Study
Arm/Group | IC51 Cohort 1 | IC51 Cohort 2 | IC51 Cohort 3
Started | 99 | 103 | 102
Enrolled and Vaccinated at Day 0 | 98 | 103 | 102
Completed | 96 | 100 | 97
Not Completed | 3 | 3 | 5
Not completed — Lost to Follow-up | 2 | 1 | 5
Not completed — Not vaccinated at Day 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Subject missed Visit 4 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IC51 Cohort 1 | IC51 Cohort 2 | IC51 Cohort 3 | Total
Number analyzed (Participants) | 98 | 103 | 102 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.3 (7.6) | 28.6 (10.7) | 31.6 (10.7) | 29.2 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 55 | 51 | 167
  Male | 37 | 48 | 51 | 136
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/ White | 93 | 98 | 102 | 293
  Asian | 5 | 5 | 0 | 10
  Black or African American | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary: 1. Geometric Mean Titers (GMT) at Day 56
Time Frame: 56 days post 1st vaccination
Population: Intention To Treat Population, i.e., all subjects entered into the study who received at least one dose of study medication
Measure: Geometric Mean (95% Confidence Interval); unit: Geometric Mean Titer - Estimate
Arm/Group | IC51 Cohort 1 | IC51 Cohort 2 | IC51 Cohort 3
Number analyzed (Participants) | 98 | 103 | 102
Geometric Mean Titer - Estimate | 100.1 [78.9 to 127.0] | 84.7 [66.3 to 108.2] | 68.1 [54.4 to 85.4]

2. Secondary Outcome: Secondary: 1. Seroconversion Rate 2. GMTs Day 28, Month 6 and Month 12 3. Treatment Emergent Adverse Events 4. Systemic and Local Tolerability
Time Frame: see above
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to Day 56
Arm/Group | IC51 Cohort 1 | IC51 Cohort 2 | IC51 Cohort 3
Serious Adverse Events (participants affected / at risk) | 2/98 | 1/103 | 0/102
Other Adverse Events (participants affected / at risk) | 66/98 | 58/103 | 61/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Cohort 1 (N=98) | IC51 Cohort 2 (N=103) | IC51 Cohort 3 (N=102)
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IC51 Cohort 1 (N=98) | IC51 Cohort 2 (N=103) | IC51 Cohort 3 (N=102)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 2
Ocular Hyperaemia (Eye disorders) | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3
Dry Mouth (Gastrointestinal disorders) | 0 | 2 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 5 | 7
Toothache (Gastrointestinal disorders) | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 3 | 20 | 10
Influenza Like Illness (General disorders) | 13 | 10 | 15
Injection Site Erythema (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 2 | 1
Cystitis (Infections and infestations) | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 3 | 0 | 2
Nasopharyngitis (Infections and infestations) | 11 | 7 | 7
Rhinitis (Infections and infestations) | 5 | 1 | 2
Sinusitis (Infections and infestations) | 1 | 1 | 1
Subcutaneous Abscess (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 2
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0
Iron Deficiency (Investigations) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 9 | 9
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Disturbance In Attention (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 3 | 2
Headache (Nervous system disorders) | 26 | 24 | 32
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Endometrial Hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Endometriosis (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other